CLINICAL TRIAL: NCT01665222
Title: Single Dose Two-Way Crossover Fasted Bioequivalence Study of Morphine Sulfate 60 mg Extended-Release Tablets in Healthy Volunteers.
Brief Title: Bioequivalence Study of Morphine Sulfate 60 mg Extended-Release Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ranbaxy Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AAI-US-456
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine Sulfate 60mg Extended-release tablets (Experimental): A single oral dose of Morphine Sulfate 60mg Extended-release tablets of Ohm Laboratories Inc.
  Interventions: Drug: Morphine Sulfate
- MS Contin® 60 mg Controlled-release tablets (Active Comparator): A single oral dose of MS Contin® 60 mg Controlled-release tablets of Purdue Pharma L.P.
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Morphine Sulfate — Morphine Sulfate 60mg Extended-release tablets

SUMMARY:
The study was to evaluate the relative bioavailability of morphine and morphine-6-glucuronide from 2 tablet products and determine if the 2 products were bioequivalent to each other.

DETAILED DESCRIPTION:
This was a single center, single-dose, randomized, open-label, two-treatment, two-period crossover bioequivalence study designed to evaluate the pharmacokinetics and bioequivalence of morphine sulfate formulations under fasted conditions. Normal healthy males and females at least 18 years of age were screened for enrollment into the trial.

Potential subjects who met the eligibility criteria randomly received either oral Morphine Sulfate 60 mg Extended-release tablets or oral MS Contin® 60 mg Controlled-release tablets on Day 1 in Period 1, then, following the washout period, they were dosed on Day 8 in Period 2 with the other treatment. There was a 7-day washout period between dosing. The study drug treatments were administered after almost a 12-hour fast. Fasting continued until slightly over 4 hours post-dose for both treatment groups. All enrolled subjects were administered single oral doses of 50 mg of naltrexone hydrochloride 10 hours predose, 1 hour predose, and 12 hours post-dose of the study drug treatment on Day -1 and Day 1 in Period 1 and on Day 7 and Day 8 in Period 2.

Potential subjects (ie, alternates) were administered single oral doses of 50 mg of naltrexone hydrochloride 10 hours predose and 1 hour predose of the study drug treatment on Day -1 and Day 1 in Period 1. Subjects visited the clinic at AAIPharma at Screening (within 28 days prior to dosing) to assess eligibility and returned to the clinic on Day -1 for the Period 1 confinement period that lasted through Day 2. To complete Period 1, subjects were to return on Day 3 for the collection of pharmacokinetic blood samples. Period 1 dosing was followed by the 7-day washout period. Subjects returned to the clinic for the Period 2 confinement period on Day 7, which continued through Day 9. To complete Period 2, subjects were to return on Day 10 in that period for the collection of pharmacokinetic and safety blood samples.

Pharmacokinetic and safety assessments were performed during the conduct of the trial. Blood samples for the evaluation of morphine and morphine-6-glucuronide plasma concentrations were obtained while subjects were at the clinic and after discharge, as appropriate. Pharmacokinetic samples were collected over a 48-hour period of time following administration of the study drug treatment.

Medical care of the subjects was assured by the presence of a physician for at least 4 hours post-dose, and the physician remained on-call to treat adverse events (AEs). Professional medical personnel were on-site during the entire study confinement period. Adverse event information elicited during Confinement at the clinic or during telephone contacts was reviewed and documented.

ELIGIBILITY:
Inclusion Criteria:

For inclusion into the trial, subjects were required to fulfill all of the following criteria:

1. Healthy subjects at least 18 years of age.
2. Willingness to provide written informed consent after being informed of the nature of the study.
3. Body mass index (BMI) between 18 and 30 and a weight of at least 110 pounds.
4. Good health as determined by a lack of clinically significant abnormalities in health assessments performed at Screening, as judged by the physician.

Exclusion Criteria:

Any of the following was regarding as a criterion for excluding subjects from the trial:

1. Hypersensitivity to morphine sulfate (MS Contin®), naltrexone (ReVia®), or related compounds.
2. Conditions that affected the absorption, metabolism, or passage of drugs out of the body (eg, sprue, celiac disease, Crohn's disease, colitis, liver, kidney, or thyroid conditions).
3. Recent history (within 1 year) of mental illness, drug addiction, drug abuse, or alcoholism.
4. A hematocrit value of ≤ 33.0% for females and ≤ 37.0% for males.
5. Donation of > 500 mL of blood in the past 8 weeks prior to study drug dosing or difficulty in donating blood.
6. Receipt of an investigational drug within the 4 weeks prior to study drug dosing.
7. Current use of any systemic prescription medications, except for oral/cutaneous/vaginal/injectable hormone contraceptives, within the 7 days prior to study drug dosing or over-the-counter (OTC) medication within 3 days of study drug dosing. This prohibition did not include vitamins or herbal preparations taken as nutritional supplements for non-therapeutic indications, as judged by the attending physician. Any nonprescription medication consumption reported was to be reviewed by the investigator prior to dosing. At the discretion of the investigator, these volunteers could be enrolled if the medication was not anticipated to alter study integrity or the safety of the subject.
8. Regular smoking of more than 5 cigarettes weekly or the regular daily use of nicotine containing products beginning 3 months before study drug administration through the final evaluation. Subjects had to be able to refrain from smoking while confined in the clinic.
9. Female subjects who were lactating or had a positive pregnancy test at Screening and prior to each of the treatment periods. Females were to use a medically acceptable method of contraception throughout the entire study period and for 1 week after study completion. Medically acceptable methods of contraception that could have been used by the subject and/or her partner were oral contraceptives/patches, progestin injection or implants, condom with spermicide, diaphragm with spermicide, intrauterine device (IUD), vaginal spermicidal or hormonal suppository, surgical sterilization of themselves or their partner(s), or abstinence. Females using contraceptive medications/devices must have used them consistently for at least 3 months prior to receiving study drug.
10. Alcohol, grapefruit beverages or foods, caffeine, or xanthine beverages or foods beginning 48 hours before each study drug administration through the last pharmacokinetic (PK) sample of each treatment period.

    Such restricted items included coffee, tea, iced tea, Coke®, Pepsi®, Mountain Dew®, chocolate, brownies, etc.
11. Regular use of any drugs known to induce or inhibit hepatic drug metabolism (examples include barbiturates, carbamazepine, rifampin, phenylhydantoins, phenothiazines, cimetidine, omeprazole, macrolides, imidazoles, fluoroquinolones) within 30 days prior to study drug administration.
12. Positive test results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), and hepatitis C antibody at Screening.
13. Positive test results for drugs of abuse or pregnancy at Screening and prior to each study drug dosing period.
14. Subjects having emesis after either dose of naltrexone administered prior to the study drug were not to be continued in the study.

Ages: 20 Years to 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2006-10; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetics | predose and at 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.333, 3.667, 4, 5, 6, 8, 10, and 12 hours post-dose
  Cmax, Area Under Curve and Tmax

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html